CLINICAL TRIAL: NCT02732535
Title: The Natural Killer Cells Regulatory Role Against Hepatic Fibrosis Following Bariatric Surgery
Brief Title: Natural Killer (NK) Cells Following Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0298-15-HMO-CTIL
Record Dates: First submitted 2015-12-02; First posted 2016-04-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2015-10

CONDITIONS: Natural Killer Cell Deficiency, Familial Isolated
MeSH Terms: conditions — Natural Killer Cell Deficiency, Familial Isolated | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: sleeve gastrectomy , roux-en-y gastric bypass — laparoscopic sleeve gastrectomy or laparoscopic gastric bypass

SUMMARY:
This study will determine the role of the NK cells before and after bariatric surgery. The investigators selected patients with NAFLD.

A Fibroscan evaluation will be assessed as a new modality to evaluate liver fibrosis.

DETAILED DESCRIPTION:
All morbidly obese patients who are candidates for a bariatric procedure in the investigators institution who has a fatty liver in their routine preoperative US will undergo a fibroscan to assess the degree of liver fibrosis preoperatively in addition to a blood sample that will be withdrawn from those participants to isolate the NK cells and to assess their activities by the assessment of the active form of NK cells (CD107a) using the spectrometry (FACS) analysis.

The investigators will also collect other clinical data including comorbidities (hypertension, diabetes mellitus and hyperlipidemia) in addition to the following routine blood test( complete blood count, creatinine, urea, International normalized ratio, liver function test, HBa1C, cholesterol, HDL, LDL, triglycerides, vitamin D, vitamin B12, potassium, sodium, albumin, bilirubin, C- reactive protein, iron, ferritin and transferrin).

All of the above mentioned tests including the NK cells and the fibroscan will be examined for all participants in 3, 6, 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* age from 18-65
* body mass index above 30 with comorbidity or above 35 with or without comorbidity
* evidence of hepatic fibrosis in routine preoperative US

Exclusion Criteria:

* patient with known other liver disease such as autoimmune or alcoholic hepatitis
* patient that take hepatotoxic medication or hormonal treatment
* active alcohol abuse above 20 gram per day
* Drug abuse
* patient refusal
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: obese patient with BMI above 30 with comorbidity or BMI above 35 with or without comorbidity, that have evidence of hepatic fibrosis on the routine preoperative US
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Determine Natural Killer (NK) cell phenotype and alterations prior and following Bariatric surgery | 1 year
  NK cells are through to play role in modulating fibrogenesis. They exert an anti-fibrotic effects by Killing activated hepatic stellate Cells; the major cells responsible for fibrosis.
  NK cells activations are crucial step in inhibiting liver fibrosis. Therefore, their functions are thought to be affected in Obese patients.
  Our aim is to investigate changes in peripheral Blood NK cells by detecting their cytotoxicity potentials by CD107a (LAMP-1; Lysosomal-associated membrane protein 1) as a marker for activation and analyze them by flow-cytometry.
  Peripheral Blood NK cells will be obtained from obese patients prior to Bariatric surgery and following 3 months, 6 months and 12 months of the surgery.

SECONDARY OUTCOMES:
To assess the fibrosis downstaging by fibroscan prior and following Bariatric surgery | 1 year
  The liver fibrosis can be assess by fibroscan and scored from 0 to 4 . all the participants will be assessed by fibroscan prior an 3,6,12 month postoperative to determine the degree of down staging of liver fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Abed Khalaileh, MD, PhD, Principal Investigator — israel ministrty of health
Locations (1):
- Hadassah Medical Organization,Jerusalem,Israel, Jerusalem, Israel, Israel

IPD SHARING:
Plan to Share IPD: Undecided